CLINICAL TRIAL: NCT01689662
Title: A Multi-center Clinical Study to Evaluate the Safety and Efficacy of FolateScan (Technetium Tc 99m EC20) in Subjects With Suspected Metastatic Renal Cell Carcinoma
Brief Title: Safety and Efficacy of FolateScan (Technetium Tc 99m EC20) in Subjects With Suspected Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC20.3
Record Dates: First submitted 2012-09-09; First posted 2012-09-21 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2012-09

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

ARMS (1):
- Tc 99m EC20 (Experimental): Subjects will receive two intravenous injections 1-3 minutes apart:
  1. 1 mg of folic acid
  2. 1-2 mL injection of 0.1 mg of EC20 labeled with 15-25 mCi of technetium-99m
  Interventions: Drug: Tc 99m EC20

INTERVENTIONS:
Drug: Tc 99m EC20

SUMMARY:
The folate receptor (FR) is overexpressed by many different cancer types, including renal cell carcinoma. Besides helping in the diagnosis of cancer, a folate-targeted imaging agent could provide an effective method to identify folate receptor-positive (FR+) cancer patients that may benefit from folate-targeted therapy. Up to 40 subjects, with known or strongly suspected metastatic renal cell carcinoma with at least one target lesion detected by a diagnostic imaging procedure (e.g. ultrasonography, CT, or MRI), will be enrolled in this study.

DETAILED DESCRIPTION:
The investigational new drug (FolateScan or Technetium Tc 99m EC20) is a folate-targeted diagnostic radiopharmaceutical designed to bind to the folate receptor. The folate receptor is a glycoprotein that is over-expressed in many types of cancer cells but it is only minimally distributed in normal tissues. Folate conjugates bind to the folate receptor with high affinity and are brought into the cell via endocytosis. In contrast, folic acid itself enters most normal cells via the reduced folate carrier, a pathway entirely inaccessible to folate conjugates. Therefore, these folate conjugates are specific to cancer cells.

Endocyte's folate-targeted delivery system was applied towards the targeting of a diagnostic imaging agent (111In-DTPA-Folate) to ovarian cancer tumors. This proof-of-principle study was designed to demonstrate the ability of folate to target drugs to folate-receptor-positive (FR+) cancer tissue.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following eligibility requirements to be enrolled in the study.

  1. Subject must be 18 years of age or older.
  2. Subject must have known or strongly suspected metastatic renal cell carcinoma with at least one target lesion as identified by ultrasonography, MRI, or CT.
  3. Subject must have good kidney function.
  4. Subject must provide written informed consent prior to enrollment.

Exclusion Criteria:

* Subjects must be excluded if any of the following conditions are present:

  1. Subject is pregnant or breastfeeding.
  2. Subject is simultaneously participating in another investigational drug study, excluding the follow-up phase.
  3. Subject has received an investigational agent within 7 days prior to enrollment.
  4. Subject is unable to tolerate conditions for radionuclide imaging.
  5. Subject has been administered another radiopharmaceutical that would interfere with the assessment of Technetium Tc 99m EC20.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-08; Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States